CLINICAL TRIAL: NCT01376258
Title: Benefits of Adherence to 5-alpha Reductase Inhibitor Treatment in Men With Enlarged Prostate: An Assessment of Medicare and Medicaid Patients Using the MarketScan Database
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113907
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Prostatic Hyperplasia
Keywords: benign prostatic hyperplasia; acute urinary retention; adherence; 5-alpha reductase inhibitor; enlarged prostate; surgery
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Finasteride; Dutasteride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients adherent to 5-alpha reductase inhibitor (5ARI): Patients with benign prostate hyperplasia (BPH) who are adherent (as measured by a medication possession ratio (MPR)) based on 3 MPR threshold values of 70%, 75% and 80%
  Interventions: Drug: 5ARI
- Patients who are non-adherent to 5ARI therapy: Patients with BPH who are not adherent to 5ARI therapy as measured by 3 MPR threshold values of 70%, 75%, and 80%
  Interventions: Drug: 5ARI

INTERVENTIONS:
Drug: 5ARI — dutasteride or finasteride
  Other Names: Proscar® (finasteride); Avodart® (dutasteride)

SUMMARY:
Adherence and length of treatment with a 5-alpha reductase inhibitor (5ARI) therapy may be associated with improved clinical outcomes for patients with enlarged prostates (EP) and lower health care related costs.

The objectives of this study are to quantify 1.) the relationship between 5ARI adherence and length of therapy and the likelihood of acute urinary retention (AUR), prostate-related surgery (emergency and non-emergency), and clinical progression (defined as AUR and/or prostate-related surgery); and 2.) the monthly EP-related, medical costs in a Medicaid and Medicare population. The null hypothesis is that no differences will be observed in the outcomes and costs of patients who adhere to long-term 5ARI therapy and those who do not. The test hypothesis is that patients with higher levels of adherence to 5ARI for a longer period of time will experience significantly fewer adverse outcomes and significantly lower treatment costs.

The data source for this analysis is the MarketScan database, which contains medical and pharmacy claims for commercial health plan members and Medicare recipients. Medical and pharmacy claims data are sourced directly from health plans and employers. The database represents approximately 18 to 20 million individuals annually and nearly 22 million Medicaid enrollees from multiple states. The database includes the Medicare-covered portion of payment, the employer-paid portion, and any out-of-pocket expenses paid by the beneficiary.

The study design is a retrospective cohort analysis. Each patient's index date was defined as the date of the first fill for a 5ARI prescription.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 65 or older
* A diagnostic claim of BPH (ICD-9-CM code 222.2x or 600.xx)
* A prescription claim for a 5ARI for at least 60 days during the observation period
* Continuous eligibility for 6 months prior to and at least 91 days after the index date

Exclusion Criteria:

* A prostate cancer diagnosis
* A procedure cost for any prostate-related surgical procedure prior to the index date

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study will include retrospective data from male patients aged 65 years and older with continuous health plan enrollment from July 1, 2003 and June 30, 2009. Patient records will be reviewed for data from the 6-months prior to and 1-year following the index date, which represents the first prescription fill for a 5ARI
Sampling Method: Non-Probability Sample
Enrollment: 28903 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Mean number of patients with a diagnosis code for acute urinary retention (AUR) and/or a procedure code for prostate surgery | 1 year following the first therapy date or until an event that signifies clinical progression is observed (whichever occurs first)
  AUR and prostate surgery are indicative of clinical progression of enlarged prostate (EP)

SECONDARY OUTCOMES:
Adjusted benign prostatic hyperplasia (BPH)-related costs | 1 year following the first therapy date
  Differences in cost will be compared across cohorts. BPH-related costs include those associated with ICD-9-CM codes 222.2x or 600.xx
Medication Possession Ratio (MPR) | 1 year following the first therapy date
  A measure of medication adherence (compliance and discontinuation) in patients taking monotherapy versus early combination therapy. Discontinuation is defined as a 30-day gap in therapy

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline